CLINICAL TRIAL: NCT01601808
Title: A Prospective, Phase II, Double Blinded, Multicentre, Randomised Clinical Trial Comparing Combination Gemcitabine and Vandetanib Therapy With Gemcitabine Therapy Alone in Locally Advanced or Metastatic Pancreatic Carcinoma
Brief Title: Clinical Trial Comparing Gemcitabine and Vandetanib Therapy With Gemcitabine Alone in Pancreatic Carcinoma
Acronym: ViP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-021951-26; 74555382 (Other: ISRCTN)
Record Dates: First submitted 2012-02-22; First posted 2012-05-18 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2012-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — vandetanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine and Placebo (Placebo Comparator): Standard therapeutic arm. Placebo orally once a day continuously together with gemcitabine 1000mg/m2 weekly as a 30 minute infusion for 7 consecutive weeks. This will then be followed by a one week break and then gemcitabine 1000mg/m2 weekly as a 30 minute infusion for 3 weeks followed by a one week break in subsequent cycles.
  Interventions: Drug: Placebo
- Gemcitabine and vandetanib (Experimental): Experimental arm. Vandetanib orally once a day continuously together with gemcitabine 1000mg/m2 weekly as a 30 minute infusion for 7 consecutive weeks. This will then be followed by a one week break and then gemcitabine 1000mg/m2 weekly as a 30 minute infusion for 3 weeks followed by a one week break in subsequent cycles.
  Interventions: Drug: Caprelsa (vandetanib)

INTERVENTIONS:
Drug: Placebo — Orally once a day, continuously throughout the study
  Arms: Gemcitabine and Placebo
Drug: Caprelsa (vandetanib) — Orally once a daily, continuously throughout the study.
  Arms: Gemcitabine and vandetanib

SUMMARY:
ViP is a double blinded clinical trial which will compare gemcitabine and vandetanib chemotherapy with gemcitabine alone in patients with locally advanced or metastatic pancreatic carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically or cytologically proven pancreatic ductal adenocarcinoma or undifferentiated carcinoma of the pancreas.
* Locally advanced or metastatic disease precluding curative surgical resection or definitive locally directed therapies such as chemo radiation. Patients who have relapsed following previously resected Pancreatic Cancer can be included.
* Contrast enhanced computerised tomography (CT) scan of the thorax, abdomen and pelvis within 28 days prior to commencing treatment.
* Unidimensionally measurable disease as shown by CT scan, in accordance with RECIST guidelines (version 1.1)
* ECOG performance status 0, 1 or 2 where the investigator feels that treatment with combination chemotherapy.
* Platelets ≥100 x 109/l; WBC ≥ 3 x 109/l; neutrophils ≥ 1.5 x 109/l at entry.
* Documented Life expectancy > 3 months.
* Informed written consent

Exclusion Criteria:

* Laboratory results:

  * Serum bilirubin ≥ 1.5x the upper limit of reference range (ULRR).
  * Haemoglobin < 10G/dl
  * Creatinine clearance < 30 mL/minute (calculated by Cockcroft-Gault formula)**. Patients with a creatinine clearance of ≥30mL/minute and <50mL/minute should begin vandetanib on a reduced dose of 200mg.
  * Potassium, ≤4.0 mmol/L despite supplementation; or > 5.5 mmol/L
  * Magnesium below the normal range despite supplementation, or > 1.23 mmol/L
  * Serum calcium is > 2.9 mmol/L. In cases where serum calcium is below the normal range this can be substituted with the value for calcium adjusted for albumin, if this is below the normal range despite supplementation patients should be excluded.
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or alkaline phosphatase (ALP) >2.5 x ULRR or > 5x ULRR if judged by the investigator to be related to liver metastases.
* Medical or psychiatric conditions compromising informed consent.
* Intracerebral metastases or meningeal carcinomatosis.
* Major surgery within 4 weeks or incompletely healed surgical incision before starting study therapy.
* Evidence of severe or uncontrolled systemic disease or any concurrent condition
* Clinically significant cardiovascular eventclassification of heart disease ≥2 within 3 months before entry; or presence of cardiac disease that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia.
* History of arrhythmia which is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled on medication is not excluded.
* QTc prolongation with other medications that required discontinuation of that medication.
* Congenital long QT syndrome or 1st degree relative with unexplained sudden death under 40 years of age.
* Presence of left bundle branch block (LBBB).
* QTc with Bazett's correction that is un-measurable or ≥ 480 msec on screening ECG. Patients who are receiving a drug that has a risk of inducing Torsades-de-Pointes are excluded if QTc is ≥ 460 msec.
* Any concurrent medication with a known risk of inducing Torsades-de-Pointes, that in the investigator's opinion cannot be discontinued, are allowed.
* Concomitant medications that are potent inducers.
* Hypertension not controlled by medical therapy.
* Currently active diarrhoea.
* Malabsorption syndrome.
* Pregnancy or breast feeding.
* Previous chemotherapy for locally advanced and metastatic disease. Adjuvant chemotherapy for resected pancreatic cancer will be permitted provided that chemotherapy was completed > 12 months previously.
* Radiotherapy within the last 4 weeks prior to start of study treatment.
* Concurrent malignancies or invasive cancers diagnosed within past 5 years.
* Chemotherapy directed at tumour apart from that described in this protocol.
* All men or women of reproductive potential, unless using at least two contraceptive precautions, one of which must be a condom.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2011-10-10 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
Overall survival | Analysis will be carried out when all patients have a minimum of 1-year follow-up after randomisation
  To assess whether survival times for patients receiving gemcitabine plus vandetanib are longer than for those patients receiving gemcitabine alone as first line treatment for advanced pancreatic cancer

SECONDARY OUTCOMES:
Progression-free survival time | Analysis will be carried out when all patients have a minimum of 1-year follow-up after randomisation
Objective response rate | Analysis will be carried out when all patients have a minimum of 1-year follow-up after randomisation
Disease control rate | Analysis will be carried out when all patients have a minimum of 1-year follow-up after randomisation
Number and types of adverse events | Analysis will be carried out when all patients have a minimum of 1-year follow-up after randomisation
Patient pain assessment | Analysis will be carried out when all patients have a minimum of 1-year follow-up after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Dr Gary Middleton, Principal Investigator — Royal Surrey County Hospital NHS Foundation Trust
Locations (14):
- United Kingdom (14):
  - Belfast City Hospital, Belfast
  - The Royal Bournemouth Hospital, Bournemouth
  - Bristol Haematology and Oncology Centre, Bristol
  - Royal Surrey County Hospital, Guildford
  - Clatterbridge Centre for Oncology, Liverpool
  - Royal Liverpool University Hospital, Liverpool
  - St Bartholomew's Hospital, London
  - Guys & St Thomas Hospital, London
  - Royal Marsden Hospital, London
  - The Christie Hospital, Manchester
  - James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle
  - Nottingham City Hospital, Nottingham
  - Weston Park Hospital, Sheffield